CLINICAL TRIAL: NCT02271646
Title: Ultrasound Guided Thoracic Paravertebral Blocks: An Effective Pain Control in Percutaneous Radiofrequency Ablation of Hepatic Tumors
Brief Title: Ultrasound Guided Thoracic Paravertebral Block for Hepatic Tumors Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 070/2557(EC2); (IO) R015731063 (Other Grant/Funding Number: Faculty of medicine, Siriraj hospital, Mahidol university)
Record Dates: First submitted 2014-09-03; First posted 2014-10-22 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Liver Cancer
Keywords: paravertebral block; ultrasound guided
MeSH Terms: conditions — Liver Neoplasms | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0.5% marcaine 20ml (Experimental): 3 levels ultrasound guided thoracic paravertebral blocks at T5-6, T7-8 and T9-10 (total 0.5% marcaine 20ml)
  Interventions: Drug: 0.5% marcaine 20ml

INTERVENTIONS:
Drug: 0.5% marcaine 20ml — 3 levels ultrasound guided thoracic paravertebral block at T5-6, T7-8 and T9-10 (total 0.5% marcaine 20ml)

SUMMARY:
Patients undergo percutaneous radiofrequency ablation of hepatic tumors at Siriraj hospital normally receive only intravenous sedative drugs which sometimes can not provide effective pain control.

TPVB is suitable for unilateral operations. And it is increasing popular nowadays because of using ultrasound guided which make it is more reliable and has less side effects especially the severe one such as pneumothorax. To cover all nerve supply liver, we decided to use right TPVB at T5-6, T7-8, and T9-10.

The aim of this study is to prove that TPVB can provide an effective pain control for patients undergo liver RFA both at rest and movement (cough). We are going to measure the pain score at recovery room and the effective pain control means patients has mild pain (pain score less </= 3 and do not ask for analgesic drugs).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients undergo percutaneous radiofrequency ablation for liver tumors
* ASA classification 1-3

Exclusion Criteria:

* Psychiatric illness
* Chronic abdominal pain > 1 week
* Regular analgesic drugs use
* Infection at back (Block area)
* Severe spinal deformity
* PT > 16 sec, aPTT > 32, platelet < 50,000/cumm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
pain score at recovery room both at rest and movement (cough) | Up to 24 hours
  All patients at recovery room has mild pain (pain score </= 3) and do not need any rescue analgesic drugs.

SECONDARY OUTCOMES:
Distribution of local anesthetic drugs after performing ultrasound guided TPVB at T5-6, T7-8 and T9-10. | After performing TPVB at 5, 10, 20 and 30 minutes.
  Test with cold sensation.

CONTACTS AND LOCATIONS:
Overall Officials: Pawinee Pangthipampai, M.D., Principal Investigator — Mahidol University
Locations (1):
- Siriraj hospital, Bangkok, Thailand